CLINICAL TRIAL: NCT06562881
Title: Patient Navigation to Improve Surgical Access in Primary Hyperparathyroidism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: American College of Surgeons (Other)
Responsible Party: Principal Investigator, Rachel Kelz, Executive Vice Chair, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 855141
Record Dates: First submitted 2024-08-12; First posted 2024-08-20 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Hyperparathyroidism, Primary
Keywords: Parathyroidectomy; Barriers and Challenges to Surgical Health Equity
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scheduling Navigation (Experimental): Participants will be assigned to a scheduler.
  Interventions: Other: Scheduling Navigation
- Without Scheduling Navigation (Active Comparator): Participants will not be assigned to a scheduler.
  Interventions: Other: Without Scheduling Navigation

INTERVENTIONS:
Other: Scheduling Navigation — Participants will be connected to a scheduler to schedule a surgical consultation visit at time of recruitment. Participation does not guarantee or require surgery.
  Arms: Scheduling Navigation
Other: Without Scheduling Navigation — Patients will work with clinic staff in the usual fashion for their treatment for primary hyperparathyroidism. They will not be connected directly to a scheduler to help schedule a surgical consultation visit at time of recruitment. With our crossover design, if patients have not yet received surgical consultation after 3 months, they will be called and connected with a scheduler at that time. Participation does not guarantee or require surgery.
  Arms: Without Scheduling Navigation

SUMMARY:
The goal of this study is to address surgical health equity in historically marginalized participants with primary hyperparathyroidism (PHPT). The main questions that this study aims to answer are, how does patient navigation impact:

* The proportion of PHPT participants undergo parathyroidectomy?
* The proportion of PHPT participants who complete surgical consultation?
* Time to surgical consultation?
* Time to surgery?

DETAILED DESCRIPTION:
Patients historically marginalized in Medicine are at increased risk of delayed care and undertreatment of PHPT, which can result in end-organ damage and reduced quality of life due to fatigue, brain fog, pain and other constitutional symptoms due to imbalances in calcium levels. It can be easily treated with a highly curative, cost-effective, and low risk surgery but less than 40% of patients who qualify for surgery undergo treatment. Patients from historically marginalized populations such as black/Hispanic/Asian race, underinsurance, and older age are disproportionately impacted by lower rates of surgery and longer delays to surgery.

This pragmatic pilot trial aims to address surgical health equity in historically marginalized patients with PHPT by assessing the impact of navigation, specifically direct outreach and appointment scheduling, on conversion of surgical referral to consultation and conversion of surgical consultation to treatment in two dimensions, timeliness and clinical outcomes. Participants will be randomized to receive or not receive scheduling navigation at time of recruitment with a crossover design at 3 months for those who do not receive scheduling navigation at time of recruitment and have yet to complete surgical consultation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PHPT and not yet had parathyroidectomy who meet criteria for surgical treatment of PHPT (osteoporosis, fragility fracture, or evidence of vertebral compression fracture on spine imaging, renal involvement [renal stone, silent nephrolithiasis on renal imaging, nephrocalcinosis, hypercalciuria (24-hour urine calcium level 400 mg/dL) with increased stone risk, or impaired renal function (glomerular filtration rate 60 mL/min)], calcium 1 mg/dL above upper limit of normal, age less than 50)
* Qualify as a member of a racial or ethnic minority group (Black, Hispanic, Asian and Pacific Islander, Native American), lower socioeconomic neighborhoods (by zipcode), socially vulnerable (social determinants of health indicating financial strain, social vulnerability index in the top quartile 75%+ by zip code), or with underinsurance (Medicaid, Medicare, dual eligible, uninsured)

Exclusion Criteria:

* Prior Parathyroidectomy
* End-stage Renal Disease
* Renal Transplant
* Vitamin D Deficiency
* Metastatic Disease
* Familial Hypocalciuric Hypercalcemia
* No Indication for Surgery
* Unable/Unwilling to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Parathyroidectomy Surgical Outcome | Within 12 months
  The primary outcome will be the proportion of patients who undergo parathyroidectomy

SECONDARY OUTCOMES:
Completion of Consultation | Through study completion, an average of 1 year after time of recruitment or surgery
  Proportion of participants who complete surgical consultation
Time to Consultation | Through study completion, an average of 1 year after time of recruitment or surgery
  Time from participant referral to scheduling and completion of surgical consultation consultation
Time to Surgery | Through study completion, an average of 1 year after time of recruitment or surgery
  Time from participant referral to surgery
Complications related to hyperparathyroidism | Assessed at 6 and 12 months after recruitment or surgery in all groups
  New, worsening, or recurrent end organ disease (osteoporosis, kidney stone, renal impairment, mental health disorders or cognitive function (requiring hospitalization or loss of independence), pancreatitis)
Parathyroidectomy complications | Assessed at 6 and 12 months after recruitment or surgery in all groups
  Complications rates of the following:
  Bleeding/hematoma Hypocalcemia Surgical site infection Voice dysfunction Tracheostomy
Persistent hyperparathyroidism | Assessed at 6 and 12 months after recruitment or surgery in all groups
  Rate of persistent disease, based on pattern of calcium and parathyroid hormone levels postoperatively
Recurrent hyperparathyroidism | Assessed at 6 and 12 months after recruitment or surgery in all groups
  Rate of recurrent disease, based on pattern of calcium and parathyroid hormone levels postoperatively)
Surgical parathyroid re-exploration | Assessed at 6 and 12 months after recruitment or surgery in all groups
  Rate of re-exploration for hyperparathyroidism

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Kelz, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States